CLINICAL TRIAL: NCT02865551
Title: The Rate of Urinary Retention in Women After Vaginal Delivery With Epidural Anesthesia Who Underwent Prolonged Catheterization Compared With Intermittent Catheterization During Labor.
Brief Title: Urinary Retention After Vaginal Delivery With Epidural Anesthesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Dr. Roy Lauterbach, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0141-15-RMB
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention | interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended catheterization (Experimental): Participants in which a foley catheter will be inserted adjacent to epidural anesthesia during labor.
  Interventions: Device: Foley catheter; Drug: Epidural anesthesia
- Intermittent catheterization (Experimental): Participants in which a short term catheter will be inserted every 4 hours during labor after epidural anesthesia until delivery.
  Interventions: Device: Short term catheter; Drug: Epidural anesthesia

INTERVENTIONS:
Device: Foley catheter — Extended bladder catheterization after epidural anesthesia.
  Arms: Extended catheterization
Device: Short term catheter — Intermittent catheterization every 4 hours after epidural anesthesia.
  Arms: Intermittent catheterization
Drug: Epidural anesthesia — Performance of epidural anesthesia by a certified anesthesiologist.

SUMMARY:
The investigators intend to compare the rate of urinary retention among female patients after vaginal delivery under epidural anesthesia, depending on bladder catheterization type, either by a foley catheter inserted adjacent to epidural anesthesia or intermittent catheterization applied every 4 hours during labor.

DETAILED DESCRIPTION:
An explanation about the study will be delivered to each participant and each participant will sign a confirmed consent. Patients will be randomized between 2 groups of treatment: 1. intermittent catheterization applied every 4 hours during labor. 2. foley catheter inserted adjacent to epidural anesthesia.

In patients with a foley catheter, the catheter will be removed soon after delivery. Participants will be followed by a clinician post labor. An abdominal US will be performed either 4 hours after delivery or after the participant urinates to check the bladder volume.

Patient information including demographic information, information regarding the patient's pregnancy and delivery will be collected from the patient's electronic record.

ELIGIBILITY:
Inclusion Criteria:

* Female patients in labor designated for vaginal delivery with epidural anesthesia.

Exclusion Criteria:

* Patients with neurological problems including gestational diabetes.
* Patients either designated for elective cesarean delivery or emergent cesarean delivery.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of urinary retention after vaginal delivery with epidural anesthesia | Up to 3 days

SECONDARY OUTCOMES:
Rate of urinary tract infections | Up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Lior Lowenstein, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No